CLINICAL TRIAL: NCT00551096
Title: A Phase I Study of Gemcitabine, Capecitabine and ZD6474 (ZACTIMA) in Patients With Advanced Solid Tumors With an Expanded Cohort of Patients With Biliary or Pancreatic Malignancies.
Brief Title: Gemcitabine/Capecitabine/ZD6474 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0129.cc
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Malignant Solid Tumour; Biliary Cancer; Pancreatic Cancer
Keywords: Advanced Solid Tumors; Biliary or Pancreatic Malignancies
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, capecitabine and ZD6474 (Experimental): Gemcitabine administered intravenously over 30 minutes on days 1, 8 and 15 of each cycle at a fixed dose of 1000mg/m2.
  Capecitabine administered orally at 1660 mg/m2/day divided into two doses for 21 days followed by a week-off .
  ZD6474 administered orally at 300 mg/day once daily. One cycle will consist of 28 days.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine; Drug: ZD6474

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine administered intravenously over 30 minutes on days 1, 8 and 15 of each cycle at a fixed dose of 1000mg/m2.
  Other Names: Gemzar
Drug: Capecitabine — Capecitabine administered orally at 1660 mg/m2/day divided into two doses for 21 days followed by a week-off.
  Other Names: Xeloda
Drug: ZD6474 — Administered orally at 300 mg/day once daily. One cycle will consist of 28 days
  Other Names: Zactima

SUMMARY:
Zactima will be used in this study to determine the highest dose that can be given safely as well as the side effects of Zactima when in combination with two FDA approved drugs; gemcitabine and capecitabine. This combination will be given to patients with advanced solid tumors. Once the highest dose of the combination has been determined, additional patients with biliary cancers (cholangiocarcinomas and gallbladder cancer) and locally advanced or metastatic pancreatic cancer will be treated at the highest determined dose for further studies.

DETAILED DESCRIPTION:
This phase I study will access a novel regimen using a multi-targeted anti-angiogenic agent which targets the tyrosine kinase of vascular endothelial growth factor (VEGF) receptor 2 and epidermal growth factor receptor (EGFR) in combination with cytotoxic agents: gemcitabine and capecitabine. The rationale is based on observations that there is an additive / synergistic effect when cytotoxic agents are combined with angiogenesis inhibitors. There is also evidence that EGFR mediated signaling pathways are potent stimulators of VEGF production. Also the concept of dual targeting of tumor and endothelial cells may provide more encouraging results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (measure of your ability to perform everyday tasks)
* Life expectancy of at least three months

Blood samples and other testing may apply for further testing of eligibility.

Exclusion Criteria:

* Uncontrolled illness (for example, current infections or heart conditions)
* Abnormal laboratory tests (such as blood or urine testing)
* Pregnant or breastfeeding women

Further exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ZACTIMA (ZD6474) in combination with Gemcitabine and Capecitabine | Up to 28 days
  To evaluate the safety profile and determine the MTD dose of ZACTIMA in combination with Gemcitabine and Capecitabine in patients with advanced malignancies. Toxicity will be graded per Common Toxicity Criteria for Adverse Effects (CTCAE) Version 3.0 and adverse event reporting for this study will be performed via Adverse Event Expedited Reporting System (AdEERS). All patients who receive any amount of the study drug will be evaluable for toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Leong, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kessler ER, Eckhardt SG, Pitts TM, Bradshaw-Pierce EL, O'byrant CL, Messersmith WA, Nallapreddy S, Weekes C, Spratlin J, Lieu CH, Kane MA, Eppers S, Freas E, Leong S. Phase I trial of vandetanib in combination with gemcitabine and capecitabine in patients with advanced solid tumors with an expanded cohort in pancreatic and biliary cancers. Invest New Drugs. 2016 Apr;34(2):176-83. doi: 10.1007/s10637-015-0316-5. Epub 2015 Dec 30. PMID 26715573